CLINICAL TRIAL: NCT06629038
Title: A Novel Technique for Estimating Maximal Jaw Movement, Neck and Shoulder Joint Range of Motion Using an Artificial Intelligence Model
Brief Title: Estimating Jaw, Neck, and Shoulder Range of Motion Using an AI Model
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202403103RINA
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Oral Cancer
Keywords: oral cancer; shoulder; range of motion; artificial intelligence; pose estimation; maximal mouth opening
MeSH Terms: conditions — Mouth Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oral cancer patients: oral cancer patients with trismus, neck, or shoulder problems
  Interventions: Behavioral: observation alone
- healthy adults: healthy adults without history of trismus, neck, or shoulder problems
  Interventions: Behavioral: observation alone

INTERVENTIONS:
Behavioral: observation alone — observation of maximal mouth opening, lateral excursion, and range of motion of shoulder abduction, neck joint

SUMMARY:
This observational study aims to develop an AI-based system for tracking mandibular and shoulder movements using deep learning techniques. It will compare AI-generated pose estimations with gold standard measurements to assess accuracy, particularly in patients with functional impairments from oral cancer treatment, such as trismus, spinal accessory nerve dysfunction, neck dystonia, and radiation fibrosis.

DETAILED DESCRIPTION:
Due to the involvement of various structures, patients with oral cancer may experience functional impairments after treatment, such as trismus, spinal accessory nerve dysfunction, neck dystonia, radiation fibrosis, and fatigue. This observational study aims to develop an AI-based system for tracking mandibular and shoulder movements using deep learning techniques. AI-generated pose estimations will be compared with gold standard measurements: maximal mouth opening will be compared with caliper measurements, and Therabilte scale, while shoulder abduction range of motion will be compared with universal goniometer measurements. We will recruit 20 healthy adults and 20 oral cancer patients. Data on maximal mouth opening and shoulder abduction will be collected through video recordings, calipers, Therabilte scale, and universal goniometers. The videos will be analyzed using deep learning to estimate mouth opening and shoulder abduction angles. These estimates will then be compared with the gold standard measurements. The Intraclass Correlation Coefficient (ICC), Mean Absolute Error (MAE), and Coefficient of Variation (CV) will be used as performance indicators to assess and compare the reliability, accuracy, and consistency of the models.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults without a history of head, neck or shoulder injury or surgery, and without HNC-related radiotherapy or chemoradiotherapy
* Oral cancer patients with trismus, clinical signs of neck or shoulder joint impairment after oral cancer surgery or radiotherapy
* Age between 20 and 65 years

Exclusion Criteria:

* Could not communicate
* Had any disorder that could influence movement performance

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community, university
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
maximal mouth opening | The date of enrollment
  maximal mouth opening
maximal lateral excursion of mandible | The date of enrollment
  maximal lateral excursion of mandible
range of motion of shoulder abduction | The date of enrollment
  range of motion of shoulder abduction
range of motion of neck | The date of enrollment
  lateral side bending and rotation of the neck

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badiola-Bengoa A, Mendez-Zorrilla A. A Systematic Review of the Application of Camera-Based Human Pose Estimation in the Field of Sport and Physical Exercise. Sensors (Basel). 2021 Sep 7;21(18):5996. doi: 10.3390/s21185996. PMID 34577204
- [Background] Sandler ML, Lazarus CL, Ru M, Sharif KF, Yue LE, Griffin MJ, Likhterov I, Chai RL, Buchbinder D, Urken ML, Ganz C. Effects of jaw exercise intervention timing on outcomes following oral and oropharyngeal cancer surgery: Pilot study. Head Neck. 2019 Nov;41(11):3806-3817. doi: 10.1002/hed.25908. Epub 2019 Aug 12. PMID 31407421
- [Background] van der Geer SJ, Reintsema H, Kamstra JI, Roodenburg JLN, Dijkstra PU. The use of stretching devices for treatment of trismus in head and neck cancer patients: a randomized controlled trial. Support Care Cancer. 2020 Jan;28(1):9-11. doi: 10.1007/s00520-019-05075-7. Epub 2019 Nov 7. PMID 31701267
- [Background] Shao CH, Chiang CC, Huang TW. Exercise therapy for cancer treatment-induced trismus in patients with head and neck cancer: A systematic review and meta-analysis of randomized controlled trials. Radiother Oncol. 2020 Oct;151:249-255. doi: 10.1016/j.radonc.2020.08.024. Epub 2020 Sep 3. PMID 32890607
- [Background] Cohen EE, LaMonte SJ, Erb NL, Beckman KL, Sadeghi N, Hutcheson KA, Stubblefield MD, Abbott DM, Fisher PS, Stein KD, Lyman GH, Pratt-Chapman ML. American Cancer Society Head and Neck Cancer Survivorship Care Guideline. CA Cancer J Clin. 2016 May;66(3):203-39. doi: 10.3322/caac.21343. Epub 2016 Mar 22. PMID 27002678
- [Background] Watters AL, Cope S, Keller MN, Padilla M, Enciso R. Prevalence of trismus in patients with head and neck cancer: A systematic review with meta-analysis. Head Neck. 2019 Sep;41(9):3408-3421. doi: 10.1002/hed.25836. Epub 2019 Jun 19. PMID 31215723
- [Background] Stenum J, Cherry-Allen KM, Pyles CO, Reetzke RD, Vignos MF, Roemmich RT. Applications of Pose Estimation in Human Health and Performance across the Lifespan. Sensors (Basel). 2021 Nov 3;21(21):7315. doi: 10.3390/s21217315. PMID 34770620
- [Background] Chen YH, Liang WA, Lin CR, Huang CY. A randomized controlled trial of scapular exercises with electromyography biofeedback in oral cancer patients with accessory nerve dysfunction. Support Care Cancer. 2022 Oct;30(10):8241-8250. doi: 10.1007/s00520-022-07263-4. Epub 2022 Jul 11. PMID 35821447
- [Background] Chen YH, Lin CR, Liang WA, Huang CY. Motor control integrated into muscle strengthening exercises has more effects on scapular muscle activities and joint range of motion before initiation of radiotherapy in oral cancer survivors with neck dissection: A randomized controlled trial. PLoS One. 2020 Aug 6;15(8):e0237133. doi: 10.1371/journal.pone.0237133. eCollection 2020. PMID 32760097
- [Background] Chen YH, Huang CY, Liang WA, Lin CR, Chao YH. Effects of Conscious Control of Scapular Orientation in Oral Cancer Survivors With Scapular Dyskinesis: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211040827. doi: 10.1177/15347354211040827. PMID 34412536
- [Background] Beshara P, Chen JF, Read AC, Lagadec P, Wang T, Walsh WR. The Reliability and Validity of Wearable Inertial Sensors Coupled with the Microsoft Kinect to Measure Shoulder Range-of-Motion. Sensors (Basel). 2020 Dec 17;20(24):7238. doi: 10.3390/s20247238. PMID 33348775
- [Background] Shepherd J, Hansjee S, Divall P, Raval P, Singh HP. How do digital range of motion measurement devices 'measure-up' to traditional goniometry in assessing shoulder range of motion? A systematic review and meta-analysis. Shoulder Elbow. 2024 Jul;16(4):363-381. doi: 10.1177/17585732231195554. Epub 2023 Aug 31. PMID 39318409
- [Background] Takigami S, Inui A, Mifune Y, Nishimoto H, Yamaura K, Kato T, Furukawa T, Tanaka S, Kusunose M, Ehara Y, Kuroda R. Estimation of Shoulder Joint Rotation Angle Using Tablet Device and Pose Estimation Artificial Intelligence Model. Sensors (Basel). 2024 May 2;24(9):2912. doi: 10.3390/s24092912. PMID 38733018
- [Background] van den Hoorn W, Lavaill M, Cutbush K, Gupta A, Kerr G. Comparison of Shoulder Range of Motion Quantified with Mobile Phone Video-Based Skeletal Tracking and 3D Motion Capture-Preliminary Study. Sensors (Basel). 2024 Jan 15;24(2):534. doi: 10.3390/s24020534. PMID 38257626